CLINICAL TRIAL: NCT06249854
Title: A Multicenter, Open Label, Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy With Bojungikki-tang and Pembrolizumab Monotherapy in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Combination Therapy With Bojungikki-tang and Pembrolizumab Monotherapy in Patients With Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, Mi-kyung Jeong, Principal researcher, Korea Institute of Oriental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIOM-NSCLC-ICT-01
Record Dates: First submitted 2024-01-09; First posted 2024-02-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Bojungikki-tang; Buzhong Yiqi decoction; Hochu-ekki-to
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Buzhong Yiqi decoction; bu-zhong-yi-qi-tang; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bojungikkitang & Pembrolizumab combination treatment group (Experimental): Pembrolizumab is administered intravenously every 3 weeks for 45 weeks according to standard procedures until disease progression (PD) or unacceptable toxicity occurs.
  Bojungikgitang is used in combination with immune checkpoint inhibitor treatment(Pembrolizumab) and is taken 1 bag twice a day before or between meals.
  Interventions: Drug: Bojungikki-tang(BJIKT); Drug: Pembrolizumab
- Pembrolizumab monotherapy group (Active Comparator): Pembrolizumab is administered intravenously every 3-week for 45 weeks according to routine practice until disease progression (PD) or unacceptable toxicity occurs.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Bojungikki-tang(BJIKT) — Bojungikgitang, which is a classical formulation widely used in South Korea, China, and Japan for a long time, has been reported to have following anticancer activities.
  1. Protective effect of intestine and hematopoietic organs against radiation damage
  2. Improving localized radiotherapy-induced immune deterioration
  3. Improving cancer-related fatigue and QOL
  4. Reducing radiation or chemotherapy induced side effects
  Other Names: Buzhong Yiqi Decoction, Hochu-ekki-to
  Arms: Bojungikkitang & Pembrolizumab combination treatment group
Drug: Pembrolizumab — It is a humanized antibody used in cancer immunotherapy for various types of cancer, including lung cancer. It targets the programmed cell death protein 1 (PD-1) receptor of lymphocytes. It was approved for medical use in the U.S. in 2014.

SUMMARY:
This is a multicenter, open-label, randomized controlled clinical trial designed to evaluate the efficacy and safety of combination therapy with Bojungikki-tang(BJIKT) and pembrolizumab monotherapy in patients with advanced non-small cell lung cancer whose tumors express PD-L1 positive with no EGFR or ALK genomic tumor aberrations.

Based on prior pre-clinical studies, the combination of Bojungikki-tang and immune checkpoint inhibitors (ICIs) can be expected to improve survival and enhance the therapeutic efficacy of ICIs by modulating the systemic tumor-immune environment.

Therefore, this clinical trial aims to assess the efficacy and safety of the combined therapy with BJIKT and pembrolizumab and establish clinical evidence for an integrative cancer treatment strategy by examining the survival rate and immune status following combined ICI and BJIKT treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized controlled clinical trial to evaluate the efficacy and safety of combination therapy with Bojungikki-tang(BJIKT) and pembrolizumab monotherapy in patients with advanced non-small cell lung cancer whose tumors express PD-L1 positive with no EGFR or ALK genomic tumor aberrations. A total of 70 patients aged 19 or older will be enrolled in the study and progression-free survival (PFS) will be assessed as the primary endpoint.

In a pre-clinical study, the combination of immune checkpoint inhibitors(ICIs) and Bojungikki-tang extended the survival of mice compared to the administration of ICIs or BJIKT alone and reduced tumor volume and weight. In addition, it was confirmed that various immune-related factors in the tumor microenvironment were controlled to improve the immunosuppressed microenvironment and to strengthen the tumor immune response by increasing major immune cytokines in the blood. Furthermore, the combination of ICIs and BJIKT did not cause pharmacodynamic and pharmacokinetic drug interactions, and significant side effects of Bojungikki-tang were not observed in most clinical reports on long-term administration of Bojungikki-tang. Based on the results, the combination of BJIKT and ICIs is expected to improve survival and enhance the therapeutic efficacy of ICIs by modulating the systemic tumor-immune environment.

In order to evaluate efficacy, variables including PFS, disease control rate (DCR), overall survival (OS), and quality of life will be used. The incidence rate of adverse events (AEs) and AEs with CTCAE grade 3 or higher will be assessed for safety. Most variables will be followed up during and after 45-week treatment, and the safety of interventions will be monitored consistently. Immune profiling and multi-omics analyses, including transcriptomic, proteomic, and metabolomic evaluations of PBMCs, will be conducted for exploratory purposes. In addition, pattern identification, a traditional diagnostic method in East Asian medicine, will be utilized as an exploratory variable. A validated questionnaire assessing Cold-Heat patterns, tongue diagnosis data, and pulse diagnosis data will be used to investigate their correlation with clinical and laboratory data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily decided to participate and provided written consent, after listening and understanding the detailed explanation about the clinical trial
2. Adult male or female aged 19 years or older
3. Patients with histologically or cytologically confirmed advanced (stage IV) non-small cell lung cancer [according to TNM 8th edition] In case of recurrence, only extra-thoracic metastasis is allowed.
4. Patients planned for immune checkpoint inhibitor (Pembrolizumab) monotherapy as first-line treatment (Patients with PD-L1 tumor proportion score(TPS) ≥ 50% and no EGFR or ALK genomic tumor aberrations)
5. Life expectancy ≥ 3 months
6. ECOG (Eastern Cooperative Oncology Group) Performance Status score of 0~2
7. Patients with at least 1 measurable lesion as defined in RECIST V1.1
8. Patients with adequate bone marrow reserve or organ function as follows:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500/㎕
   * Platelet count ≥100× 10^3/㎕
   * Serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 45 ml/min (measured using standard methods at the study site)
   * ALT and AST ≤ 2.5× ULN Patients with liver metastasis: ALT and AST ≤ 5× ULN
   * Total bilirubin ≤ 1.5× ULN Patients with liver metastasis or known Gilbert syndrome(unconjugated hyperbilirubinemia): Total bilirubin ≤ 3× ULN

Exclusion Criteria:

1. Active brain metastases accompanied by clinically significant neurological symptoms or signs
2. Patients who diagnosed with another primary malignancy that affect non-small cell lung cancer in the last 5 years However, effectively treated non-melanoma skin cancer, carcinoma in situ of cervix, ductal carcinoma in situ of breast, thyroid cancer, or malignancies which were remained in remission during more than 3 years after being treated effectively and considered cured are permitted.
3. Patients who treated with immune checkpoint inhibitor or anti-CTLA-4 within the last 6 weeks or systemic immunosuppressive medications within the last 2 weeks However, low-dose corticosteroids (prednisone ≤ 10 mg/day or an equivalent dose of corticosteroid within 7 consecutive days) are permitted at the investigator's discretion.
4. Patients receiving thiazide or loop diuretics
5. Hypokalemia (less than 3.0 mEq/L)
6. Active interstitial lung disease requiring oral or intravenous steroid treatment
7. Patients with autoimmune disease requiring systemic treatment at the time of enrollment
8. Uncontrolled diabetes mellitus at the time of enrollment (Uncontrolled with insulin and oral medications, HbA1c ≥ 8.0% or fasting blood sugar ≥ 200 mg/dL)
9. Patients with uncontrolled hypertension at the time of enrollment (systolic pressure > 150 mmHg or diastolic pressure >100 mmHg) despite use of antihypertensive agent
10. Patients with uncontrolled heart disease (severe heart failure, unstable angina, uncontrolled arrhythmia, or history of life-threatening arrhythmia, etc.)
11. Patients with hereditary problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, etc.
12. Patient with known active or uncontrolled HIV, tuberculosis, hepatitis B, or hepatitis C infection
13. Pregnant or lactating women
14. Patients who do not agree to use effective contraception during treatment period and for at least 5 months after the end of IP administration
15. Patients who received herbal medicine within 4 weeks before the first administration of IP (Bojungikgitang) and been decided that such intake affect the trial or safety of the subject at the investigator's discretion
16. Patients who received other investigational drugs within 30 days before the first administration of IP (Bojungikgitang)
17. Severe hypersensitivity to IP and its components (rash, redness, hives, eczema, dermatitis, itching, etc.)
18. Patients who are not eligible for the trial at the discretion of the investigator including severe infectious diseases or organ failure, etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Every 9 weeks until PD(progressive disease), up to end of study (2 years from study initiation)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Every 9 weeks until PD(progressive disease), up to end of study (2 years from study initiation)
Overall Survival (OS) | Upon confirmation of death, end of the study (2 years from study initiation)
Object Response Rate (ORR) | Every 9 weeks until PD(progressive disease), up to end of study (2 years from study initiation)
Time to Progression (TTP) | Every 9 weeks until PD(progressive disease), up to end of study (2 years from study initiation)
Duration of Response (DoR) | End of study (2 years from study initiation)
Time to Treatment Failure (TTF) | Every 9 weeks until PD(progressive disease), up to end of study (2 years from study initiation)
Number of participants with hyper-progressive disease | Up to end of study (2 years from study initiation)
Quality of Life (QoL) | Baseline, Visit 4(week 10), End of Treatment(EOT) visit(week 46)
Correlation between immuno/omics data and clinical data | Baseline, week 4, week 10, week 19, week 28, week 37, End of Treatment(EOT) visit(week 46)
Treatment response according to classification of the cold-heat pattern | End of study (2 years from study initiation)
  Cold-heat pattern classification (Cold pattern, Non-cold pattern, Heat pattern, Non-heat) refers to pattern identification of traditional East Asian medicine diagnosed by experts (Doctors of Korean Medicine) based on validated questionnaire, digital tongue diagnosis system data, and digital pulse diagnosis system data
Pulse waveform analysis of digital pulse diagnostic system | Baseline, Visit 4(week 10), End of Treatment(EOT) visit(week 46)
  The Electric Radial Tonometry device complies with ISO 18615:2020.
Data of digital tongue diagnosis system | Baseline, Visit 4(week 10), End of Treatment(EOT) visit(week 46)
  Categorical scales including tongue colors of tongue body: pale, light pink, red, and continuous variables including the Commission Internationale del'Éclairage (CIE) L*a*b* color values of tongue that represent the brightness, saturation of red and green, and saturation of blue and yellow, respectively.
  The equipment used in this study has an algorithm to increase repeatability and diagnostic accuracy by using indirect illumination and feedback gridlines. Also, it was designed to meet the international standards ISO 20498-1, 20498-2, 20498-3, 20498-4, and 20498-5.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Lee, Ph.D, Principal Investigator — Koera University Guro Hospital
Locations (7):
- South Korea (7):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Kyung Hee University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Samsung medical center, Seoul
  - Korea University Guro Hospital, Seoul
  - The catholic university of Korea Seoul Saint. Mary's hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pai-Scherf L, Blumenthal GM, Li H, Subramaniam S, Mishra-Kalyani PS, He K, Zhao H, Yu J, Paciga M, Goldberg KB, McKee AE, Keegan P, Pazdur R. FDA Approval Summary: Pembrolizumab for Treatment of Metastatic Non-Small Cell Lung Cancer: First-Line Therapy and Beyond. Oncologist. 2017 Nov;22(11):1392-1399. doi: 10.1634/theoncologist.2017-0078. Epub 2017 Aug 23. PMID 28835513
- [Background] Postow MA, Sidlow R, Hellmann MD. Immune-Related Adverse Events Associated with Immune Checkpoint Blockade. N Engl J Med. 2018 Jan 11;378(2):158-168. doi: 10.1056/NEJMra1703481. No abstract available. PMID 29320654
- [Background] Sharma P, Hu-Lieskovan S, Wargo JA, Ribas A. Primary, Adaptive, and Acquired Resistance to Cancer Immunotherapy. Cell. 2017 Feb 9;168(4):707-723. doi: 10.1016/j.cell.2017.01.017. PMID 28187290
- [Background] Pishvar M, Amirkhosravi M, Altan MC. Magnet Assisted Composite Manufacturing: A Flexible New Technique for Achieving High Consolidation Pressure in Vacuum Bag/Lay-Up Processes. J Vis Exp. 2018 May 17;(135):57254. doi: 10.3791/57254. PMID 29863655
- [Background] Kimura M, Sasada T, Kanai M, Kawai Y, Yoshida Y, Hayashi E, Iwata S, Takabayashi A. Preventive effect of a traditional herbal medicine, Hochu-ekki-to, on immunosuppression induced by surgical stress. Surg Today. 2008;38(4):316-22. doi: 10.1007/s00595-007-3631-4. Epub 2008 Mar 27. PMID 18368320
- [Background] Peng M, Li X, Lei G, Weng YM, Hu MX, Song QB. The efficacy and safety of immune checkpoint inhibitor combination therapy in lung cancer: a systematic review and meta-analysis. Onco Targets Ther. 2018 Oct 24;11:7369-7383. doi: 10.2147/OTT.S177318. eCollection 2018. PMID 30425525
- [Background] Qi F, Zhao L, Zhou A, Zhang B, Li A, Wang Z, Han J. The advantages of using traditional Chinese medicine as an adjunctive therapy in the whole course of cancer treatment instead of only terminal stage of cancer. Biosci Trends. 2015 Feb;9(1):16-34. doi: 10.5582/bst.2015.01019. PMID 25787906